CLINICAL TRIAL: NCT02132468
Title: A Ph 2 Study to Investigate the Safety and Activity of Fosbretabulin Tromethamine (CA4P) in the Treatment of Well-Differentiated, Low-to-Intermediate-Grade Unresectable, Recurrent or Metastatic PNET or GI-NET Neuroendocrine Tumors/Carcinoid With Elevated Biomarkers
Brief Title: A Ph 2 Study of Fosbretabulin in Subjects w Pancreatic or Gastrointestinal Neuroendocrine Tumors w Elevated Biomarkers
Acronym: GI-NETorPNET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX4218s
Record Dates: First submitted 2014-05-02; First posted 2014-05-07 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Neuroendocrine Tumors
Keywords: PNET; GI-NET; neuroendocrine; carcinoid
MeSH Terms: conditions — Neuroendocrine Tumors; Neuroectodermal Tumors, Primitive; Carcinoid Tumor | interventions — fosbretabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fosbretabulin tromethamine (Experimental): Fosbretabulin 90 mg/vial; 60 mg/m2, IV infusion over 10 minutes; 1x/wk; three 3-week cycles
  Interventions: Drug: fosbretabulin tromethamine

INTERVENTIONS:
Drug: fosbretabulin tromethamine — 60 mg/m2, IV on Day 1, 8 and 15 of a 3-week cycle; 3 cycles or until progression or unacceptable toxicity
  Other Names: fosbretabulin, combretastatin A4-phosphate, CA4P

SUMMARY:
This study will investigate the safety, symptoms and biomarker response of subjects with biopsy-proven well-differentiated, low-to-intermediate-grade, unresectable, or metastatic pancreatic neuroendocrine tumors (PNETs) or or Gastrointestinal Neuroendocrine tumors (GI-NETs) with elevated biochemical markers who have relapsed during or after receiving prior standard of care therapies, including octreotide, chemotherapy or targeted therapy.

DETAILED DESCRIPTION:
Subjects enrolled in this PNET/GI-NET study (OX4218s) will receive weekly dosing with fosbretabulin for up to 3 cycles or approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read, understand and provide written consent to participate in the study
* Age ≥ 18 years
* Biopsy-proven well-differentiated, low-to-intermediate-grade PNET or GI-NET with elevated (> ULN) biomarkers (serotonin, 5-hydroxyindoleacetic acid (5-HIAA), chromogranin A (CgA), neurokinin A, and neuron-specific enolase (NSE))
* Life expectancy > 12 weeks
* Must have received or may still be receiving one or more therapies including octreotide or serotonin synthesis inhibitor (SSI) or other somatostatin analogues
* Confirmed progressive disease within 18 months of enrollment on study
* Recovered from prior radiation therapy or surgery
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/µL (without growth factors)
* Platelet count ≥ 100,000/µL
* Adequate renal function as evidenced by serum creatinine

  ≤ 2.0 mg/dL (177 µmol/L)
* Adequate hepatic function: serum total bilirubin ≤ 2X greater than the upper limit of normal (ULN) (≤ 3X ULN in subjects with liver metastases), aspartate aminotransferase) AST) / alanine aminotransferase (AST) ≤ 2X the ULN for the local reference lab (≤ 5X the ULN for subjects with liver metastases)
* Disease that can be assessed (evaluable) with imaging (CT, MRI, PET, radionuclide imaging or other imaging modality)
* Women of childbearing potential as well as fertile men and their partners must use an effective method of birth control

Exclusion Criteria:

* Inadequately controlled hypertension defined as BP > 150/100 mm Hg despite medication
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Recent history (within 6 months of start of screening) of unstable angina pectoris pattern, myocardial infarction (including non-Q wave MI), or NYHA (New York Heart Association) Class III and IV Congestive Heart Failure (CHF)
* Subjects who have clinical evidence of carcinoid-induced heart disease
* History of prior cerebrovascular accident (CVA), including transient ischemic attach (TIA)
* Known central nervous system (CNS) disease except for treated brain metastasis
* History of torsade de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (<60 bpm), heart block (excluding 1st degree block, being PR interval prolongation only), congenital long QT syndrome or new ST segment elevation or depression or new Q wave on ECG
* Corrected QT interval (QTc) > 480 msec
* Ongoing treatment with any drugs known to prolong the QTc interval, including anti-arrhythmic medications (stable regimen of antidepressants of the selective serotonin reuptake inhibitor (SSRI) class is allowed))
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Significant vascular disease or recent peripheral arterial thrombosis
* Known intolerance of or hypersensitivity to fosbretabulin
* History of solid organ transplant or bone marrow transplant
* Any other intercurrent medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* High grade or poorly differentiated NET
* NET tumor other than PNET or GI-NET
* No elevated biomarker (>ULN) that can be followed
* Received regional hepatic infusion therapy within 6 months of enrollment (RFA allowed >6 months prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - Markey Cancer Center, Clinical Research Office, Lexington, Kentucky
  - Montefiore, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Froedtert Hospital, Medicial College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fosbretabulin Tromethamine
Started | 18
Completed | 11
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Fosbretabulin Tromethamine
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved, Stable, or Worsened Change In Chromogranin A (CgA) Biomarker Levels From Baseline
Description: The mean change from baseline in chromogranin A (CgA) biomarker level is considered improved if a 25% reduction occurs and worsened if the mean change from baseline is increased by 25%.
Time Frame: Baseline and 4 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine
Number analyzed (Participants) | 18
Participants
  Improved | 1
  Stable | 11
  Worsened | 6

2. Primary Outcome: Number of Participants With Improved, Stable, or Worsened Change In 5-hydroxyindoleacetic Acid (5-HIAA) Biomarker Levels From Baseline
Description: The mean change from baseline in 5-hydroxyindoleacetic acid (5-HIAA) biomarker level is considered improved if a 25% reduction occurs and worsened if the mean change from baseline is increased by 25%.
Time Frame: Baseline and 4 months
Population: Participants who had 5-hydroxyindoleacetic acid (5-HIAA) biomaker sample taken at baseline and at 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine
Number analyzed (Participants) | 13
Participants
  Improved | 2
  Stable | 8
  Worsened | 3

3. Primary Outcome: Number of Participants With Improved, Stable, or Worsened Change In Serotonin Biomarker Levels From Baseline
Description: The mean change from baseline in serotonin biomarker level is considered improved if a 25% reduction occurs and worsened if the mean change from baseline is increased by 25%.
Time Frame: Baseline and 4 months
Population: Participants who had serotonin biomaker samples taken at baseline and at 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine
Number analyzed (Participants) | 12
Participants
  Improved | 0
  Stable | 10
  Worsened | 2

4. Secondary Outcome: Number of Participants With Partial Response (PR), Progressive Disease (PD), or Stable Disease (SD) Based on RECIST 1.1
Description: The objective response rate (complete response, partial response, progressive disease, or stable disease) was determined by the investigator assessment of the participant's CT or MRI using Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1) for target lesions. Partial Response (PR) is when there is at least 30% decrease in sum of the longest diameter of the target lesions. Progressive Disease (PD) is when there is at least 20% increase in the sum of the longest diameter of the target lesions, as well as an absolute increase of at least 5 mm (including appearance of new lesions). Stable Disease (SD) is when there neither a PR nor PD is noted.
Time Frame: Baseline and 4 months
Population: Modified Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fosbretabulin Tromethamine
Number analyzed (Participants) | 14
Participants
  Partial Response | 1
  Stable Disease | 7
  Progressive Disease | 6

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Fosbretabulin Tromethamine
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fosbretabulin Tromethamine (N=18)
Carcinoid Syndrome (Endocrine disorders) | 1
Pneumonia (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fosbretabulin Tromethamine (N=18)
Anaemia (Blood and lymphatic system disorders) | 4
Leukaemoid reaction (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Carcinoid Syndrome (Endocrine disorders) | 1
Conjunctivitis Allergic (Eye disorders) | 1
Macular fibrosis (Eye disorders) | 1
vision blurred (Eye disorders) | 1
abdominal discomfort (Gastrointestinal disorders) | 1
abdominal distension (Gastrointestinal disorders) | 1
abdominal pain (Gastrointestinal disorders) | 7
abdominal pain upper (Gastrointestinal disorders) | 1
anal pruritus (Gastrointestinal disorders) | 1
ascites (Gastrointestinal disorders) | 1
constipation (Gastrointestinal disorders) | 3
diarrhoea (Gastrointestinal disorders) | 4
dyspepsia (Gastrointestinal disorders) | 1
epigastric discomfort (Gastrointestinal disorders) | 1
flatulence (Gastrointestinal disorders) | 2
eructation (Gastrointestinal disorders) | 1
frequent bowel movements (Gastrointestinal disorders) | 2
gastrointestinal pain (Gastrointestinal disorders) | 1
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
hypoaesthesia oral (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 6
vomiting (Gastrointestinal disorders) | 4
breakthrough pain (General disorders) | 1
chest pain (General disorders) | 2
chills (General disorders) | 3
early satiety (General disorders) | 1
fatigue (General disorders) | 11
feeling jittery (General disorders) | 1
injection site bruising (General disorders) | 1
local swelling (General disorders) | 1
non-cardiac chest pain (General disorders) | 1
oedema peripheral (General disorders) | 4
pyrexia (General disorders) | 4
hepatic failure (Hepatobiliary disorders) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
upper respiratory tract infection (Infections and infestations) | 1
urinary tract infection (Infections and infestations) | 5
urosepsis (Infections and infestations) | 1
infusion related reaction (Injury, poisoning and procedural complications) | 3
upper limb fracture (Injury, poisoning and procedural complications) | 1
alanine aminotransferase increased (Investigations) | 6
aspartate aminotransferase increased (Investigations) | 6
blood alkaline phosphatase increased (Investigations) | 3
blood creatinine increased (Investigations) | 1
blood magnesium increased (Investigations) | 1
weight decreased (Investigations) | 1
white blood cell count increased (Investigations) | 1
decreased appetite (Metabolism and nutrition disorders) | 3
dehydration (Metabolism and nutrition disorders) | 2
diabetes mellitus (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
hyperkalaemia (Metabolism and nutrition disorders) | 1
hypoalbuminaemia (Metabolism and nutrition disorders) | 3
hypocalcaemia (Metabolism and nutrition disorders) | 1
hypokalaemia (Metabolism and nutrition disorders) | 3
hypomagnesaemia (Metabolism and nutrition disorders) | 3
hypophosphataemia (Metabolism and nutrition disorders) | 1
hypovolaemia (Metabolism and nutrition disorders) | 1
metabolic acidosis (Metabolism and nutrition disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 7
bone pain (Musculoskeletal and connective tissue disorders) | 2
connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1
flank pain (Musculoskeletal and connective tissue disorders) | 3
muscle spasms (Musculoskeletal and connective tissue disorders) | 1
muscular weakness (Musculoskeletal and connective tissue disorders) | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
myalgia (Musculoskeletal and connective tissue disorders) | 1
neck pain (Musculoskeletal and connective tissue disorders) | 2
pain in jaw (Musculoskeletal and connective tissue disorders) | 1
cranial nerve disorder (Nervous system disorders) | 1
dizziness (Nervous system disorders) | 1
encephalopathy (Nervous system disorders) | 1
headache (Nervous system disorders) | 3
migraine (Nervous system disorders) | 1
neuralgia (Nervous system disorders) | 1
neuropathy peripheral (Nervous system disorders) | 3
paraesthesia (Nervous system disorders) | 4
restless leg syndrome (Nervous system disorders) | 2
tremor (Nervous system disorders) | 1
anxiety (Psychiatric disorders) | 1
depression (Psychiatric disorders) | 1
dysuria (Renal and urinary disorders) | 1
polyuria (Renal and urinary disorders) | 1
proteinuria (Renal and urinary disorders) | 1
renal failure (Renal and urinary disorders) | 1
renal failure acute (Renal and urinary disorders) | 1
urinary retention (Renal and urinary disorders) | 1
prostatitis (Reproductive system and breast disorders) | 1
pruritis genital (Reproductive system and breast disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 2
dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
blister (Skin and subcutaneous tissue disorders) | 1
hyperhydrosis (Skin and subcutaneous tissue disorders) | 1
night sweats (Skin and subcutaneous tissue disorders) | 5
pruritis (Skin and subcutaneous tissue disorders) | 5
pruritis generalised (Skin and subcutaneous tissue disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 2
rosacea (Skin and subcutaneous tissue disorders) | 1
flushing (Vascular disorders) | 4
hypertension (Vascular disorders) | 3
hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days